CLINICAL TRIAL: NCT02391285
Title: Mitigating Chronic Pelvic Floor Dysfunction Following Childbirth by Pelvic Floor Dynamometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STH18128 V1.0, 05 April 2014
Record Dates: First submitted 2014-11-06; First posted 2015-03-18 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Pelvic Floor Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pelvic floor dynamometry (Experimental)
  Interventions: Device: dynamometer (Auckland vaginal elastometer)

INTERVENTIONS:
Device: dynamometer (Auckland vaginal elastometer) — The elastometer is a modified vaginal speculum which captures pelvic muscle tone over 3 minutes and records this on an attached computer. In addition to the elastometer test, there are three further related tests, which patients would be suitable to participate in.
  I. a questionnaire to fill in so as to obtain some feedback from patients regarding what they thought of the test and the device.
  II. The investigators would like to repeat the elastometer measurement within a week of the first test to determine the reliability and accuracy of repeating the measurement after a few days.
  III. The investigator would like to request that the patient have an MRI scan of the pelvic muscles to check whether the elastometer can pick up functional muscle weakness that would not otherwise be recognised except by performing an MRI scan. The investigators will therefore compare elastometer readings to the MRI scan findings.
  Other Names: elastometer

SUMMARY:
To assess the potential clinical utility of measuring pelvic floor muscle tone after childbirth by vaginal dynamometry, the investigators will study 50 consecutive consenting first attendees of the Jessop Wing perineal trauma clinic. In addition to clinical and imaging assessment routinely offered women at this clinic, the investigators will measure their active and passive pelvic floor muscle tone using the Auckland vaginal elastometer. The investigators will also assess structural pelvic floor muscle damage (PFMD) in a subset of 10 women (5 symptomatic and 5 asymptomatic) by Magnetic Resonance Imaging (MR) scan of the pelvic hiatus. The investigators will then determine the predictive capacity of vaginal elastometry for symptoms of pelvic floor damage, findings of endoanal sonography, and MR scans of the pelvic floor hiatus. The investigators will determine if vaginal elastometry can prove an objective and accurate frontline assessment tool for the management of PFMD following childbirth. Our observations will generate vital data for powering and designing a large clinical trial evaluating the potential use of the vaginal elastometer as a first line assessment tool of PFMD in the postnatal period. Data will also inform the design of a personalised model for predicting and managing pelvic floor muscle damage during childbirth.

DETAILED DESCRIPTION:
In recent years, vaginal dynamometry (VD) using an elastometer has emerged as a potential tool for the functional evaluation of the pelvic floor musculature, with early reports suggesting that it accurately measures and discriminates pelvic floor muscle stiffness in women of different parities, fitness levels and clinical situations including the evaluation of stress urinary incontinence (UI) [11-14].

With the emerging promising reports confirming the accuracy of the dynamometer for assessing PFM strength in various women groups and for investigating stress UI, a portable dynamometer has recently been developed by our collaborators at the Auckland Bioengineering Institute (ABI), led by Professor Poul Nielsen [15]. The device has several advantages over other designs: (1) It is hand-held, portable; (2) It is designed to be operated by a medical professional; (3) It measures in the coronal as well as the anteroposterior orientations; (4) Data acquisition is at a high frequency (100Hz) and can be automated, and (5) Parameters are adjustable to required protocols.

The device consists of a hand-piece comprising two aluminium arms, with detachable acetyl plastic speculum ends, actuated via a load cell. The tip of the speculum is wider than the neck in order to focus the measurements at the level of the puborectalis portion of the Levator Ani (LA) muscle group by reducing contributions from perineal muscles. The hand-piece is connected to a control box with a data acquisition device that communicates with a computer via a USB connection. The device measures the passive force and the displacement (i.e. speculum separation), and displays the data in a graph. The preliminary test of the portable prototype conducted in Auckland found the device highly acceptable, consistent and repeatable [15]. A recent study of 47 antenatal patients in Auckland showed 100% positive feedback for the device to be used as a regular test in the antenatal unit (internal communication).

Indicative approval has been discussed and agreed with the Department of Clinical Engineering, subject to satisfactory safety checks scheduled for March 2014, that the device is highly likely to meet safety regulatory standards for medical devices to be used on patients in the National Health Service (NHS). The device has now arrived in Sheffield and has successfully undergone safety checks in the Clinical Engineering Department of the Royal Hallamshire Hospital (certificate attached). The investigators therefore envisage that a pilot study can be carried out using the device in the Jessop Wing (JW) twice-monthly perineal trauma clinic.

The clinical studies in this setting will generate, for the first time in the United Kingdom, sensitivity and specificity data for vaginal dynamometry for detecting functional defects of PFM tone post-delivery. The Investigators will accrue data regarding the correlation of findings with clinically detected perineal muscle damage as well as radiologically-confirmed LA hiatus defects.

The success of these pilot studies will provide strong support for the investigators to seek funding for a large multicentre study of the clinical application of VD in screening and management of PFMD to prevent long term pelvic floor laxity, stress UI, and pelvic organ prolapse (POP).There is a paucity of reports regarding its application in clinical care for managing PFMD from childbirth.

The investigators will prospectively recruit 50 consecutive women attending the perineal trauma clinic (PTC) at the Jessop Wing of the Royal Hallamshire Hospital Sheffield for standard clinical care and VD. Given limitations in funding and time duration for these experiments, the investigators will adopt this pragmatic approach to recruit and study consecutive consenting women over a 6-month period.

ELIGIBILITY:
All women referred to the PTC of the JW will be eligible for inclusion in the study if they agree. Women who have had previous perineal surgery or surgery for genital prolapse or stress UI will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Stiffness Measurement (Newtons) and correlation with muscular defects on pelvic MRI and endo-anal sonography (composite measure) | 6 months
  measure pelvic floor muscle stiffness (Newtons) and validate pelvic floor muscle assessment by VD against image--based detection of anatomical deficits and damage to the levator ani and perineal muscles.
Pelvic Floor Stiffness Measurements (Newtons) and correlation with subjective clinical assessment and symptom questionnaires (EPAQPF) (composite measure) | 6 months
  measure pelvic floor muscle stiffness (Newtons) and validate pelvic floor muscle assessment by VD against subjective clinical assessment of pelvic floor tone and perineal defects, and findings from symptom assessment questionnaires and acceptability questionnaires from service users
generation of test-retest reliability data presented as a force (N) and displacement (mm) time chart and as a force---displacement X--Y plot. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jessop Wing, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No